CLINICAL TRIAL: NCT03548571
Title: Open Label Randomized Phase II/III Trial of Dendritic Cell Immunotherapy Against Cancer Stem Cells in Glioblastoma Patients Receiving Standard Therapy (DEN-STEM)
Brief Title: Dendritic Cell Immunotherapy Against Cancer Stem Cells in Glioblastoma Patients Receiving Standard Therapy
Acronym: DEN-STEM
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Einar Vik-Mo, Senior consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEN-STEM
Record Dates: First submitted 2018-04-30; First posted 2018-06-07 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Open label, randomized
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DC immunization (Experimental): Leukapheresis before start of radiotherapy. Immunization with DCs starting first week after finalizing radiotherapy (2Gy x 30) and concomitant temozolomide.
  Interventions: Biological: Dendritic cell immunization
- Standard therapy (Active Comparator): Radiotherapy (2 Gy x30) with concomitant and adjuvant temozolomide.
  Interventions: Drug: Adjuvant temozolomide

INTERVENTIONS:
Biological: Dendritic cell immunization — Intradermal injection
  Arms: DC immunization
Drug: Adjuvant temozolomide — After a 4-week break, patients were then to receive up to six cycles of adjuvant temozolomide according to the standard 5-day schedule every 28 days at 150 mg per square meter for the first cycle and thereafter increase to 200 mg per square meter beginning with the second cycle.
  Other Names: Standard therapy
  Arms: Standard therapy

SUMMARY:
Open, randomized study of a trivalent dendritic cell therapy compared to standard therapy in primary treated patients with IDH wild-type, MGMT-promotor methylated glioblastoma. The IMP is dendritic cells transfected with mRNA of survivin, hTERT og autologous tumor stem cells derived from tumorspheres.

DETAILED DESCRIPTION:
Autologous leukapheresis for enrichment of PBMCs is performed after enrollment of the patient into the trial. Ex vivo generated DCs will be frozen and stored in the vapour phase of liquid nitrogen.

At first surgery, tumor biopsies will be cultured under sphere-forming conditions under ex vivo conditions for enrichment of glioblastoma stem cells. mRNA will purified and amplified from these autologous tumor stem cells.

At specified intervals patients randomized to the vaccine group will receive intradermal injections of DCs transfected with mRNA from autologous tumor stem cells, survivin and hTERT. Injections will be given as three separate injections at three separate sites.

Vaccination will be continued for as long as there are vaccines available.

ELIGIBILITY:
Inclusion Criteria:

All of the following conditions must apply:

* Must be at least 18 years and less than 70 years of age.
* Must be ambulatory with a ECOG performance status 0 or 1
* Must have histologically confirmed glioblastoma IDH wild-type, with unmethylated MGMT-gene promotor, and a candidate for combined radiation therapy and chemotherapy ("Stupps Regimen").
* Must have accessible volume and quality of tumor tissue for vaccine production (proliferation of cells and extraction of tumor mRNA) at first surgery.
* Must have postoperative MRI after surgery with contrast enhancing tumor remnant of less than 1 cm3 or less than 10% of original tumor volume.
* Normal organ function defined by laboratory values as following: ANC > 1.5 x 109/L; platelets >100 x109/L, Hb >9g/dL (> 5.6 mmol/L). Creatinine < 140 µmol/L (1.6 mg/dL); if borderline, the creatinine clearance >40 mL/min, Bilirubin < 20% above the upper limit of normal, ASAT and ALAT < 2.5 the upper limit of normal. Albumin >2.5 g/L.
* Serology indicating contagious HIV, HBV, HCV and Treponema pallidum must be negative.
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH GCP, and national/local regulations.

Exclusion Criteria:

* Tumor in a localization where a modest increase in size due to reactive oedema may have a large impact on the patient's neurological condition, i.e. brain stem.
* History of prior malignancy other than glioblastoma, with the exception of curatively treated basal cell or squamous cell carcinoma of the skin and ca. cervicis stage IB.
* Active infection requiring antibiotic therapy.
* Significant cardiac or other medical illness that would limit activity or survival, such as severe congestive heart failure, unstable angina, or serious cardiac arrhythmia.
* Prior splenectomy.
* Glucocorticoid treatment not possible to terminate due to autoimmune disease or increased intracranial pressure.
* Adverse reactions to vaccines such as asthma, anaphylaxis or other serious reactions.
* History of immunodeficiency or autoimmune disease such as rheumatoid arthritis, systemic lupus erythematosus, scleroderma, polymyositis-dermatomyositis, juvenile onset insulin dependent diabetes, or a vasculitic syndrome.
* Chemotherapy or other potentially immune-suppressive therapy outside protocol that has been administered within the last 4 weeks prior to vaccination.
* Positive pregnancy test in women of childbearing potential (within 7 days before the first vaccination). Women of childbearing potential and sexually active male participants must use reliable methods of contraception during the whole treatment period and 3 months after the last trial drug dose. Reliable methods of contraception are defined in section .
* Any reason why, in the opinion of the investigator, the patient should not participate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-26 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 2 years
  Defined as time from first surgery to first certain progress of contrast enhancing tumor or clinical progression, according to the Response Assessment in Neuro-Oncology (RANO) criteria.

SECONDARY OUTCOMES:
Overall survival | 2 years from inclusion
  Survival from the time of diagnosis.
Patient reported quality of life, overall | 2 years from inclusion
  Evaluated by EORTC Quality of Life Questionaire (QLQ-C30), a questionnaire developed to assess the quality of life of cancer patients. Scale 30 to 120 points, where higher is worse.
Patient reported quality of life, brain specific | 2 years from inclusion
  Evaluated by EORTC Quality of Life Questionaire, Brain module (QLQ-BN20). The brain cancer module is meant for use among brain cancer patients varying in disease stage and treatment modality. Scale 20 to 80 points, where higher is worse. It should always be complemented by the QLQ-C30.
Immunological response, skin | 2 years from inclusion
  Evaluated by delayed type hypersensitivity reaction in skin.
Immunological response, cellular | 2 years from inclusion
  Evaluated by lymphocyte clonal analysis.
Adverse events | 2 years from inclusion
  Classified according to Common Terminology Criteria for Adverse Events (CTCAE).

CONTACTS AND LOCATIONS:
Overall Officials: Iver A Langmoen, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vik-Mo EO, Nyakas M, Mikkelsen BV, Moe MC, Due-Tonnesen P, Suso EM, Saeboe-Larssen S, Sandberg C, Brinchmann JE, Helseth E, Rasmussen AM, Lote K, Aamdal S, Gaudernack G, Kvalheim G, Langmoen IA. Therapeutic vaccination against autologous cancer stem cells with mRNA-transfected dendritic cells in patients with glioblastoma. Cancer Immunol Immunother. 2013 Sep;62(9):1499-509. doi: 10.1007/s00262-013-1453-3. Epub 2013 Jul 2. PMID 23817721
- [Derived] Woroniecka K, Fecci PE. Immuno-synergy? Neoantigen vaccines and checkpoint blockade in glioblastoma. Neuro Oncol. 2020 Sep 29;22(9):1233-1234. doi: 10.1093/neuonc/noaa170. No abstract available. PMID 32691060